CLINICAL TRIAL: NCT05383677
Title: ANIfrolumab Treatment for 24 Weeks in Patients With Primary Sjögren's Syndrome - Efficacy and Safety Assessment in a Randomized, Double-blind, Placebo-controlled Phase-IIa Proof-of-concept Trial (ANISE-II)
Brief Title: Anifrolumab Treatment for 24 Weeks in Patients With Primary Sjögren's Syndrome
Acronym: ANISE-II
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Medical Center Groningen (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ESR-21-21284; 2022-000609-28 (EudraCT Number)
Record Dates: First submitted 2022-03-29; First posted 2022-05-20 (Actual); Last update posted 2022-12-19 (Actual); Status verified 2022-12

CONDITIONS: Sjogren's Syndrome
MeSH Terms: conditions — Sjogren's Syndrome | interventions — anifrolumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Anifrolumab (Active Comparator): 20 patients will receive anifrolumab treatment
  Interventions: Drug: Anifrolumab
- Placebo (Placebo Comparator): 10 patients will receive placebo treatment
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Anifrolumab — Anifrolumab 300 mg will be administered in intravenous infusions once per 4 weeks, for a total treatment period of 24 weeks.
  Other Names: Saphnelo
  Arms: Anifrolumab
Drug: Placebo — Placebo will be administered in intravenous infusions once per 4 weeks, for a total treatment period of 24 weeks.
  Arms: Placebo

SUMMARY:
The ANISE-II study is a randomized, double-blind, placebo-controlled phase IIa proof-of-concept trial. Thirty patients with primary Sjögren's syndrome (pSS) are randomized in a 2:1 ratio to either anifrolumab or placebo treatment for 24 weeks. Main inclusion criteria are fulfilment of the ACR/EULAR classification criteria for pSS, disease duration of ≤10 years, and an ESSDAI and/or ESSPRI of ≥5 (at least 50% of patients need to fulfil the ESSDAI ≥5 criterion). The primary outcome measure is Composite of Relevant Endpoints for Sjögren's Syndrome (CRESS) response at week 24.

DETAILED DESCRIPTION:
The aim is to evaluate safety and determine the effects of anifrolumab on essential clinical and biological parameters in patients with primary Sjögren's syndrome (pSS). Although the pathogenesis of pSS has not been fully elucidated, one of the key immune pathways involved is type-I IFN signalling. Since anifrolumab is a fully human, IgG1κ monoclonal antibody to type-I interferon receptor subunit 1, the hypothesis is that inhibition of type-I IFN signalling by anifrolumab may reduce glandular and systemic inflammation and attenuate disease activity in patients with pSS. The study population will consist of patients who fulfil 2016 ACR-EULAR criteria for pSS and have active disease, defined by a EULAR Sjögren Syndrome Disease Activity Index (ESSDAI) score ≥5 and/or an unacceptable patient symptom state (EULAR Sjögren Syndrome Patient Reported Index (ESSPRI) score ≥5. The primary endpoint is the Composite of Relevant Endpoints for Sjögren's Syndrome (CRESS) at week 24.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent
2. Female or male aged ≥18 years
3. Disease duration (time since diagnosis) ≤10 years. In case of pediatric-onset pSS a disease duration of ≤15 years is allowed if there is residual gland function (UWS≥0.01 or SWS≥0.1 ml/min).
4. Fulfilment of 2016 ACR-EULAR classification criteria for pSS (which includes focus score ≥1 in salivary gland biopsy and/or anti-SSA/Ro positivity), based on previous diagnostic examinations
5. Presence of anti-SSA antibodies
6. ESSDAI≥5 and/or ESSPRI≥5. ESSDAI≥5 implicates a moderate to high systemic disease activity and ESSPRI≥5 implicates that the patient-reported symptom state is unacceptable. At least 50% of patients need to fulfil the ESSDAI≥5 criterion. Inclusion of patients with low ESSDAI (<5) should be discontinued when 15 included patients (50%) have a low ESSDAI.
7. Willingness to undergo a repeated parotid gland biopsy at baseline and 24 weeks after start treatment. If a recent parotid gland biopsy (within ≤1 year before the baseline visit) is available, and enough material of this parotid gland biopsy is available, this biopsy can be used as baseline sample.
8. Use of reliable method of contraception for participants of reproductive potential.
9. Vaccinated against COVID-19 (at least two COVID-19 vaccinations) or previous confirmed COVID-19 infection (from which the patient is recovered) in combination with at least one COVID-19 vaccination or a previous confirmed COVID-19 infection (from which the patients has recovered) in combination with a positive anti-SARS-CoV-2 antibody test.

Exclusion Criteria:

1. Presence of any other connective tissue disease
2. Positive pregnancy test (urinary HCG) at screening or breast-feeding
3. History of alcohol or drug abuse
4. History of malignancy or with a current suspicion for cancer, apart from local MALT lymphoma, squamous or basal cell carcinoma of the skin treated with documented success of curative therapy ≥3 months prior to week 0 or cervical cancer in situ treated with apparent success with curative therapy ≥1 year prior to week 0.
5. Subjects with evidence (as assessed by the investigator) of active or latent bacterial or viral infections at the time of potential enrollment, including subjects with evidence of HIV which will be tested during screening.
6. History of chronic or recurrent serious infections. (e.g. chronic pyelonephritis, osteomyelitis or bronchiectasis).
7. Subjects with serious bacterial infections within the last 3 months, unless treated and resolved with antibiotics.
8. Opportunistic infection requiring hospitilization or IV antimicrobial treatment within 3 years of randomization
9. Any infection requiring hospitalization or treatment with IV anti-infective medications not completed at least 4 weeks prior to signing the ICF.
10. Subjects with herpes zoster that resolved less than 12 weeks before potential enrollment or any severe case of herpes zoster in a subjects history, including, but not limited to, non-cutaneous herpes (ever), herpes encephalitis (ever), recurrent herpes zoster (defined as 2 episodes within 2 years) or ophthalmic herpes involving the retina (ever).
11. Any clinical cytomegalovirus (CMV) and Epstein-Barr virus (EBV) infection that has not completely resolved within 12 weeks prior to signing the ICF.
12. Any history of severe COVID-19 infection (e.g. requiring hospitalization, ICU care or assisted ventilation) or any prior COVID-19 infection with unresolved sequelae. Any acute COVID-19 infection (lab confirmed or suspected based on clinical symptoms) within the last 3 months prior to screening.
13. Subjects at risk for TB. Specifically excluded from this study will be subjects with a history of active TB; current clinical, radiographic, or laboratory evidence of active TB, which will be tested during screening; history of latent TB, with the exception of latent TB with documented completion of appropriate treatment.
14. Subjects who are positive for hepatitis B surface antigen, which will be tested during screening.
15. Subjects who are positive for hepatitis C antibody if the presence of hepatitis C virus was also shown with polymerase chain reaction or recombinant immunoblot assay, which will be tested during screening.
16. Subjects who have received any live or attenuated vaccines within 8 weeks prior to signing the ICF.
17. Blood transfusion or receipt of blood products within 4 weeks prior to signing the ICF.
18. Underlying cardiac, pulmonary, metabolic, renal, hepatic, gastrointestinal, hematological or neurological conditions, chronic or latent infectious diseases or immune deficiency which places the patient at an unacceptable risk for participation in the study.
19. Preceding treatment with biological DMARDs, including abatacept, anti-TNF or other monoclonal antibodies within 6 months, and rituximab within 12 months from baseline
20. Use of high-dose prednisone, less than 2 weeks before inclusion. Stable low dose (≤10 mg) is allowed.
21. Use of hydroxychloroquine, methotrexate, cyclophosphamide, cyclosporine, azathioprine, MMF and leflunomide less than 3 months ago.
22. Use of pilocarpine less than 1 month ago.
23. Lab abnormalities:

    * Serum creatinine > 2.8 mg/dl (250 μmol/l)
    * ASAT or ALAT outside 2.5 x upper normal range of the laboratory
    * Hb < 9 g/dl (5.6 mmol/l) for males and 8.5 g/dl (5.3 mmol/l) for females
    * Neutrophil granulocytes less than 0.5 x 109/l
    * Platelet count less than 50 x 109/l
24. Any other laboratory test results that, in the opinion of the investigator, might place a subject at unacceptable risk for participation in the study.
25. A known history of allergy or reaction to any component of the IP formulation or history of anaphylaxis to any human gamma globuline therapy.
26. Involvement in the planning and/or conduct of the study (applies to both Investigator staff and/or staff at the study site)
27. Previous enrolment or randomisation in the present study
28. Participation in another clinical study with an investigational drug during the last 6 months, or local investigational product during the last month

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2024-05-01 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
Composite of Relevant Endpoints for Sjögren's Syndrome (CRESS) response | Week 24
  The CRESS is a recently developed composite endpoint which consists of five clinically relevant items for pSS: a systemic disease activity, patient-reported symptoms, tear gland, salivary gland and serology item. A CRESS responder is someone who reached response on at least three out of five items (Arends et al., https://doi.org/10.1016/S2665-9913(21)00122-3)

SECONDARY OUTCOMES:
Safety (adverse events and tolerability) | Weeks 0, 4, 8, 12, 16, 20 and 24
  Adverse events and tolerability
Total CRESS response | Week 12
  The CRESS is a recently developed composite endpoint which consists of five clinically relevant items for pSS: a systemic disease activity, patient-reported symptoms, tear gland, salivary gland and serology item. A CRESS responder is someone who reached response on at least three out of five items (Arends et al., https://doi.org/10.1016/S2665-9913(21)00122-3)
ClinESSDAI | Weeks 0, 8, 12, 20, 24
  Change in ClinESSDAI from baseline, scale 0-135. A higher score means a worse outcome.
ESSPRI | Weeks 0, 8, 12, 20, 24
  Change in ESSPRI from baseline, scale 0-10. A higher score means a worse outcome.
Schirmer's test | Weeks 0, 12, 24
  Change in Schirmer's test from baseline, scale 0-35 mm. A higher score means a better outcome.
Ocular Staining Score (OSS) | Weeks 0, 12, 24.
  Change in OSS from baseline, scale 0-12. A higher score means a worse outcome
Salivary gland ultrasonography (SGUS) | SGUS: weeks 0, 12, 24
  Change in total Hocevar score (0-48) from baseline. A higher score means a worse outcome.
Rheumatoid factor (RF) | Weeks 0, 8, 12, 20, 24
  Change in RF (IU/ml) from baseline. A higher score means a worse outcome.
Total IgG | Weeks 0, 8, 12, 20, 24
  Change in IgG (g/L) from baseline. A higher score means a worse outcome.
Unstimulated whole salivary secretion (UWS) | Weeks 0, 12, 24.
  Change in UWS (reported in ml/min) from baseline. A higher score means a better outcome.
ESSDAI | Weeks 0, 8, 12, 20, 24
  Change in ESSDAI from baseline, scale 0-123. A higher score means a worse outcome.
(Clin)ESSDAI minimal clinically important improvement (MCII) | Weeks 8, 12, 20, 24
  (Clin)ESSDAI MCII is defined as a decrease of ≥3 points
(Clin)ESSDAI low disease activity | Weeks 8, 12, 20, 24
  (Clin)ESSDAI low disease activity is defined as a score<5
Physician GDA (PhGDA) | Weeks 0, 8, 12, 20, 24
  Change in PhGDA from baseline, scale 0-10. A higher score means a worse outcome.
NRS score oral, ocular and vaginal dryness | Weeks 0, 8, 12, 20, 24
  Change in NRS score from baseline, scale 0-10. A higher score means a worse outcome.
Patient GDA (PtGDA) | Weeks 0, 8, 12, 20, 24
  Change in PtGDA from baseline, scale 0-10. A higher score means a worse outcome.
Short Form-36 (SF-36) health survey | Weeks 0, 12, 24
  The SF-36 includes 8 domains, each ranging on a scale from 0-100. A higher score means a better outcome.
EurQoL 5 dimensions (EQ-5D) measure of health-related quality of life | Weeks 0, 8, 12, 20, 24
  The EQ-5D is reported as index value (0-1). A higher score means a better outcome.
Multidimensional Fatigue Index (MFI) scale | Weeks 0, 12, 24
  The MFI is reported on a scale of 4-20 for both physical and mental fatigue. A higher score means a worse outcome.
Female Sexual Function Index (FSFI) in females | Weeks 0, 12, 24
  The FSFI total score has a range of 2-36. A higher score indicates better outcome.
SGUS OMERACT score | Weeks 0, 12, 24
  The OMERACT score is reported on a scale of 0-3. A higher score means a worse outcome.
Parotid gland histology: focus score | Week 0, 24
  Number of foci / 4 mm2
Parotid gland histology: area of CD45 infiltrate | Week 0, 24
  Change in are of CD45 infiltrate at week 24 compared to week 0
Serum levels of anti-SSA/SSB | Weeks 0, 8, 12, 20, 24
  U/ml
Complement (C3/C4) | Weeks 0, 8, 12, 20, 24
  g/L
Lymphocyte count | Weeks 0, 8, 12, 20, 24
  10^9/L
Presence of cryoglobulinemia | Weeks 0, 12, 24
  Presence of cryoglobulinemia (yes/no) will be analysed at week 0, 12 and 24.

CONTACTS AND LOCATIONS:
Overall Officials: Hendrika Bootsma, Principal Investigator — University Medical Center Groningen
Locations (1):
- University Medical Centre Groningen, Groningen, Netherlands